CLINICAL TRIAL: NCT03054753
Title: Prospective Sensor Controlled Compliance Analysis of Shoulder Abduction Splint After Rotator Cuff Repair
Acronym: SENSABDUKT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Balgrist University Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: W633
Record Dates: First submitted 2017-01-31; First posted 2017-02-16 (Actual); Last update posted 2021-07-21 (Actual); Status verified 2021-07

CONDITIONS: Rotator Cuff Tear
Keywords: Abduction brace; Compliance; Rotator cuff tear; Rotator cuff repair
MeSH Terms: conditions — Rotator Cuff Injuries; Patient Compliance

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Abduction brace wearing time analysis (Other): The abduction brace wearing time analysis is performed in patients, who undergo a rotator cuff repair with postoperative abduction brace treatment
  Interventions: Behavioral: Abduction brace wearing time analysis

INTERVENTIONS:
Behavioral: Abduction brace wearing time analysis — To evaluate the patient´s abduction brace wearing time a sensor = Orthotimer® (Rollerwerk, 72336 Balingen, Germany, www.orthotimer.com) is implanted in the abduction brace. The sensor measures the body temperature of the patient. Through that the wearing time can be evaluated.

SUMMARY:
The postoperative shoulder rehabilitation in an abduction brace after rotator cuff reconstruction of the shoulder is crucial for a successful healing of the reconstruction.

In this study the investigators want to analyse the abduction brace-wearing time using a electronic sensor, which is implanted in the abduction brace. The participants will be informed about the sensor after completion of the abduction brace rehabilitation 6 weeks postoperatively.

DETAILED DESCRIPTION:
After arthroscopic reconstruction of a rotator cuff tear the healing depends on a tension free positioning of the reconstructed tendon. Therefore a abduction brace is administered routinely for 6 weeks. The re-rupture rate of rotator cuff reconstruction is about 30%. One of the reason may be mechanical overuse caused by non wearing of the abduction brace. From experience the investigators suggest that the abduction brace wearing behaviour differs among patients. The participant´s wearing compliance has been evaluated by Silverio et al. with a questionary but never with a sensor. In this study the investigators want to analyse the participant´s abduction brace wearing compliance by using an sensor, which is implanted in the abduction brace and monitors the wearing time, which reveals the objective wearing time.

The sensor is a certificated sensor, which measures temperature in °C every 15 min. If the abduction brace is worn by the participants the body temperature can be captured by the sensor. If the measured temperature is over 33°C the sensor capture the time period as a "worn" time. With this measurements the abduction brace wear time should be captured objectively. A similar kind of sensors were used to evaluate the wearing time of scoliosis-braces in patients with adolescent idiopathic scoliosis (Miller DJ eta al., Morton A et al., Takemitsu et al.) With a questionary the participants are asked of the wearing time before they will be informed about the implanted sensor. This answer represents the subjective wearing time.

The first endpoint of the study is the evaluation of the objective and subjective abduction wearing time. The second endpoint is the evaluation of the correlation between compliance and subjective outcome.

ELIGIBILITY:
Inclusion Criteria:

* Patients with rotator cuff repair and postoperative abduction for 6 weeks

Exclusion Criteria:

* Revision surgery

Min Age: 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2017-03-31 (Actual); Primary Completion 2020-12-01 (Actual); Study Completion 2021-07-01 (Actual)

PRIMARY OUTCOMES:
Objective abduction brace wearing time | 6 weeks postoperative
  A sensor is implanted in the abduction brace, which captures every 15min. the temperature. If the abduction brace is worn the sensor can measure the body temperature. The objective wearing time can be evaluated.

SECONDARY OUTCOMES:
Correlation of compliance and functional outcome | 1 year postoperative
  Compliance: Constant score:
  Compliance= objective wearing time a day in correlation to functional outcome (Shoulder Constant score 0-100pts)
Correlation of compliance and subjective outcome | 3 months postoperative
  Compliance:subjective shoulder value Compliance = objective wearing time a day in correlation to subjective shoulder value
Correlation of compliance and patient satisfaction | 3 months postoperative
  Compliance: patient satisfaction Compliance = objective wearing time a day in correlation to patient satisfaction (excellent =4, good =3, moderate=2, poor=1)

CONTACTS AND LOCATIONS:
Overall Officials: Samy Bouaichqa, MD PD, Study Chair — Balgrist University Hospital
Locations (1):
- Balgrist University Hospital, University, Zurich, Zuri, Switzerland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Silverio LM, Cheung EV. Patient adherence with postoperative restrictions after rotator cuff repair. J Shoulder Elbow Surg. 2014 Apr;23(4):508-13. doi: 10.1016/j.jse.2013.09.018. Epub 2014 Feb 24. PMID 24581418
- [Background] Miller DJ, Franzone JM, Matsumoto H, Gomez JA, Avendano J, Hyman JE, Roye DP Jr, Vitale MG. Electronic monitoring improves brace-wearing compliance in patients with adolescent idiopathic scoliosis: a randomized clinical trial. Spine (Phila Pa 1976). 2012 Apr 20;37(9):717-21. doi: 10.1097/BRS.0b013e31822f4306. PMID 22517480
- [Background] Morton A, Riddle R, Buchanan R, Katz D, Birch J. Accuracy in the prediction and estimation of adherence to bracewear before and during treatment of adolescent idiopathic scoliosis. J Pediatr Orthop. 2008 Apr-May;28(3):336-41. doi: 10.1097/BPO.0b013e318168d154. PMID 18362800
- [Background] Takemitsu M, Bowen JR, Rahman T, Glutting JJ, Scott CB. Compliance monitoring of brace treatment for patients with idiopathic scoliosis. Spine (Phila Pa 1976). 2004 Sep 15;29(18):2070-4; discussion 2074. doi: 10.1097/01.brs.0000138280.43663.7b. PMID 15371711